CLINICAL TRIAL: NCT00209339
Title: A Study of the Evalve Cardiovascular Valve Repair System Endovascular Valve Edge-to-Edge REpair STudy (EVEREST I).
Brief Title: Feasibility Study of a Percutaneous Mitral Valve Repair System.
Acronym: EVEREST(I)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Elizabeth McDermott, Divisional Vice President of Regulatory and Clinical Affairs, Abbott Vascular Structural Heart (Evalve, Inc)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol #0301; Protocol #0301
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency
Keywords: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency; Mitral Valve; MR; Mitral Valve Prolapse; E2E - Edge to Edge; Alfieri Technique; MitraClip; Functional MR; Degenerative MR; Echocardiogram; CAD - Coronary Artery Disease; Heart Failure; Heart Attack; EVEREST; EVEREST I; EVEREST II
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Coronary Artery Disease; Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MitraClip (Experimental): Percutaneous mitral valve repair (MitraClip Implant)
  Interventions: Device: Percutaneous mitral valve repair (MitraClip Implant)

INTERVENTIONS:
Device: Percutaneous mitral valve repair (MitraClip Implant) — Phase I evaluation of the safety and effectiveness of an endovascular approach to the repair of mitral valve regurgitation using the Evalve MitraClip Cardiovascular Valve Repair System.
  Other Names: EVEREST I, MitraClip

SUMMARY:
Prospective, multi-center, Phase I study of the Evalve Cardiovascular Valve Repair System (CVRS) in the treatment of mitral valve regurgitation. Patients will undergo 30-day, 6 month, 12 month, and 5 year clinical follow-up.

DETAILED DESCRIPTION:
Phase I evaluation of the safety and effectiveness of an endovascular approach to the repair of mitral valve regurgitation using the Evalve Cardiovascular Valve Repair System.

The study is a prospective, multi-center, Phase I study of the Evalve Cardiovascular Valve Repair System (CVRS) in the treatment of mitral valve regurgitation. A minimum of 20 patients will be enrolled (an additional maximum of 12 roll in-patients, a maximum of 2 per site, may be enrolled and analyzed separately). Patients will undergo 30-day, 6 month and 12 month clinical follow-up.

Up to 12 clinical sites throughout the US may participate.

The primary endpoint is acute safety at thirty days, with a secondary efficacy endpoint of reduction of MR.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe mitral regurgitation, symptomatic or asymptomatic with evidence of left ventricular dysfunction;
* Experience regurgitation origination from the central two-thirds of the valve;
* Qualify as a candidate for mitral valve surgery including cardiopulmonary bypass.

Exclusion Criteria:

* Ejection fraction < 30%
* Endocarditis
* Rheumatic heart disease
* Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-07; Primary Completion 2006-02 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Feldman, M.D., Principal Investigator — Endeavor Health
Locations (1):
- Evanston Northwestern Healthcare, Evanston, Illinois, United States

REFERENCES:
- [Background] St Goar FG, Fann JI, Komtebedde J, Foster E, Oz MC, Fogarty TJ, Feldman T, Block PC. Endovascular edge-to-edge mitral valve repair: short-term results in a porcine model. Circulation. 2003 Oct 21;108(16):1990-3. doi: 10.1161/01.CIR.0000096052.78331.CA. Epub 2003 Oct 6. PMID 14530193
- [Background] Fann JI, St Goar FG, Komtebedde J, Oz MC, Block PC, Foster E, Butany J, Feldman T, Burdon TA. Beating heart catheter-based edge-to-edge mitral valve procedure in a porcine model: efficacy and healing response. Circulation. 2004 Aug 24;110(8):988-93. doi: 10.1161/01.CIR.0000139855.12616.15. Epub 2004 Aug 9. PMID 15302782
- [Background] Herrmann HC, Rohatgi S, Wasserman HS, Block P, Gray W, Hamilton A, Zunamon A, Homma S, Di Tullio MR, Kraybill K, Merlino J, Martin R, Rodriguez L, Stewart WJ, Whitlow P, Wiegers SE, Silvestry FE, Foster E, Feldman T. Mitral valve hemodynamic effects of percutaneous edge-to-edge repair with the MitraClip device for mitral regurgitation. Catheter Cardiovasc Interv. 2006 Dec;68(6):821-8. doi: 10.1002/ccd.20917. PMID 17080467
- [Background] Silvestry FE, Rodriguez LL, Herrmann HC, Rohatgi S, Weiss SJ, Stewart WJ, Homma S, Goyal N, Pulerwitz T, Zunamon A, Hamilton A, Merlino J, Martin R, Krabill K, Block PC, Whitlow P, Tuzcu EM, Kapadia S, Gray WA, Reisman M, Wasserman H, Schwartz A, Foster E, Feldman T, Wiegers SE. Echocardiographic guidance and assessment of percutaneous repair for mitral regurgitation with the Evalve MitraClip: lessons learned from EVEREST I. J Am Soc Echocardiogr. 2007 Oct;20(10):1131-40. doi: 10.1016/j.echo.2007.02.003. Epub 2007 Jun 13. PMID 17570634
- [Background] Luk A, Butany J, Ahn E, Fann JI, St Goar F, Thornton T, McDermott L, Madayag C, Komtebedde J. Mitral repair with the Evalve MitraClip device: histopathologic findings in the porcine model. Cardiovasc Pathol. 2009 Sep-Oct;18(5):279-85. doi: 10.1016/j.carpath.2008.07.001. Epub 2008 Aug 13. PMID 18703359
- [Background] Herrmann HC, Kar S, Siegel R, Fail P, Loghin C, Lim S, Hahn R, Rogers JH, Bommer WJ, Wang A, Berke A, Lerakis S, Kramer P, Wong SC, Foster E, Glower D, Feldman T; EVEREST Investigators. Effect of percutaneous mitral repair with the MitraClip device on mitral valve area and gradient. EuroIntervention. 2009 Jan;4(4):437-42. doi: 10.4244/eijv4i4a76. PMID 19284064
- [Background] Rogers JH, Yeo KK, Carroll JD, Cleveland J, Reece TB, Gillinov AM, Rodriguez L, Whitlow P, Woo YJ, Herrmann HC, Young JN. Late surgical mitral valve repair after percutaneous repair with the MitraClip system. J Card Surg. 2009 Nov-Dec;24(6):677-81. doi: 10.1111/j.1540-8191.2009.00901.x. Epub 2009 Jul 24. PMID 19682161
- [Background] Argenziano M, Skipper E, Heimansohn D, Letsou GV, Woo YJ, Kron I, Alexander J, Cleveland J, Kong B, Davidson M, Vassiliades T, Krieger K, Sako E, Tibi P, Galloway A, Foster E, Feldman T, Glower D; EVEREST Investigators. Surgical revision after percutaneous mitral repair with the MitraClip device. Ann Thorac Surg. 2010 Jan;89(1):72-80; discussion p 80. doi: 10.1016/j.athoracsur.2009.08.063. PMID 20103209
- [Background] Franzen O, Baldus S, Rudolph V, Meyer S, Knap M, Koschyk D, Treede H, Barmeyer A, Schofer J, Costard-Jackle A, Schluter M, Reichenspurner H, Meinertz T. Acute outcomes of MitraClip therapy for mitral regurgitation in high-surgical-risk patients: emphasis on adverse valve morphology and severe left ventricular dysfunction. Eur Heart J. 2010 Jun;31(11):1373-81. doi: 10.1093/eurheartj/ehq050. Epub 2010 Mar 10. PMID 20219746
- [Background] Tamburino C, Ussia GP, Maisano F, Capodanno D, La Canna G, Scandura S, Colombo A, Giacomini A, Michev I, Mangiafico S, Cammalleri V, Barbanti M, Alfieri O. Percutaneous mitral valve repair with the MitraClip system: acute results from a real world setting. Eur Heart J. 2010 Jun;31(11):1382-9. doi: 10.1093/eurheartj/ehq051. Epub 2010 Mar 18. PMID 20299349
- [Background] Ussia GP, Barbanti M, Tamburino C. Feasibility of percutaneous transcatheter mitral valve repair with the MitraClip system using conscious sedation. Catheter Cardiovasc Interv. 2010 Jun 1;75(7):1137-40. doi: 10.1002/ccd.22415. PMID 20336809
- [Background] Jonsson A, Settergren M. MitraClip catheter-based mitral valve repair system. Expert Rev Med Devices. 2010 Jul;7(4):439-47. doi: 10.1586/erd.10.23. PMID 20583881
- [Background] Mauri L, Garg P, Massaro JM, Foster E, Glower D, Mehoudar P, Powell F, Komtebedde J, McDermott E, Feldman T. The EVEREST II Trial: design and rationale for a randomized study of the evalve mitraclip system compared with mitral valve surgery for mitral regurgitation. Am Heart J. 2010 Jul;160(1):23-9. doi: 10.1016/j.ahj.2010.04.009. PMID 20598968
- [Background] Geidel S, Ostermeyer J, Lass M, Schmoeckel M. Complex surgical valve repair after failed percutaneous mitral intervention using the MitraClip device. Ann Thorac Surg. 2010 Jul;90(1):277-9. doi: 10.1016/j.athoracsur.2009.12.048. PMID 20609795
- [Background] Kalarus Z, Kukulski T, Lekston A, Streb W, Sikora J, Nadziakiewicz P, Gasior M, Polonski L, Zembala M. [Methodology and safety of transvascular reduction of severe ischaemic mitral insufficiency with MitraClip in high-surgical-risk patients - first three cases in Poland]. Kardiol Pol. 2010 Jun;68(6):729-35. Polish. PMID 20806217
- [Background] Lim DS, Kunjummen BJ, Smalling R. Mitral valve repair with the MitraClip device after prior surgical mitral annuloplasty. Catheter Cardiovasc Interv. 2010 Sep 1;76(3):455-9. doi: 10.1002/ccd.22547. PMID 20839359
- [Background] Ciobanu A, Bennett S, Azam M, Clark A, Vinereanu D. Incremental value of three-dimensional transoesophageal echocardiography for guiding double percutaneous MitraClip (R) implantation in a 'no option' patient. Eur J Echocardiogr. 2011 Feb;12(2):E11. doi: 10.1093/ejechocard/jeq118. Epub 2010 Sep 27. PMID 20876188
- [Background] Tamburino C, Imme S, Barbanti M, Mule M, Pistritto AM, Aruta P, Cammalleri V, Scarabelli M, Mangiafico S, Scandura S, Ussia GP. Reduction of mitral valve regurgitation with Mitraclip(R) percutaneous system. Minerva Cardioangiol. 2010 Oct;58(5):589-98. PMID 20948505
- [Background] Borgia F, Di Mario C, Franzen O. Adenosine-induced asystole to facilitate MitraClip placement in a patient with adverse mitral valve morphology. Heart. 2011 May;97(10):864. doi: 10.1136/hrt.2010.208132. Epub 2010 Oct 29. No abstract available. PMID 21036802
- [Result] Feldman T, Kar S, Rinaldi M, Fail P, Hermiller J, Smalling R, Whitlow PL, Gray W, Low R, Herrmann HC, Lim S, Foster E, Glower D; EVEREST Investigators. Percutaneous mitral repair with the MitraClip system: safety and midterm durability in the initial EVEREST (Endovascular Valve Edge-to-Edge REpair Study) cohort. J Am Coll Cardiol. 2009 Aug 18;54(8):686-94. doi: 10.1016/j.jacc.2009.03.077. PMID 19679246
- [Derived] Foster E, Kwan D, Feldman T, Weissman NJ, Grayburn PA, Schwartz A, Rogers JH, Kar S, Rinaldi MJ, Fail PS, Hermiller J, Whitlow PL, Herrmann HC, Lim DS, Glower DD; EVEREST Investigators. Percutaneous mitral valve repair in the initial EVEREST cohort: evidence of reverse left ventricular remodeling. Circ Cardiovasc Imaging. 2013 Jul;6(4):522-30. doi: 10.1161/CIRCIMAGING.112.000098. Epub 2013 Apr 30. PMID 23633132
- [Derived] Siegel RJ, Biner S, Rafique AM, Rinaldi M, Lim S, Fail P, Hermiller J, Smalling R, Whitlow PL, Herrmann HC, Foster E, Feldman T, Glower D, Kar S; EVEREST Investigators. The acute hemodynamic effects of MitraClip therapy. J Am Coll Cardiol. 2011 Apr 19;57(16):1658-65. doi: 10.1016/j.jacc.2010.11.043. PMID 21492763
- [Derived] Ladich E, Michaels MB, Jones RM, McDermott E, Coleman L, Komtebedde J, Glower D, Argenziano M, Feldman T, Nakano M, Virmani R; Endovascular Valve Edge-to-Edge Repair Study (EVEREST) Investigators. Pathological healing response of explanted MitraClip devices. Circulation. 2011 Apr 5;123(13):1418-27. doi: 10.1161/CIRCULATIONAHA.110.978130. Epub 2011 Mar 21. PMID 21422390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 55 EVEREST I patients were enrolled at 11 sites.The first EVEREST I patient was enrolled on July 2, 2003 and the last patient was enrolled on February 15, 2006.
Pre-assignment Details: Patients with moderate-to-severe (3+) or severe (4+) mitral regurgitation determined from a transthoracic echocardiogram (TTE), who were candidates for mitral valve (MV) surgery and cardiopulmonary bypass were considered for enrollment in this study.
Period: At 12 Months Follow-up
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Started | 55
Completed | 40
Not Completed | 15
Not completed — Withdrawal by Subject | 8
Not completed — Death | 1
Not completed — No MitraClip Device Implanted | 6
Period: At 24 Months Follow-up
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Started | 40
Completed | 29
Not Completed | 11
Not completed — Withdrawal by Subject | 4
Not completed — Withdrawal because of other reasons | 6
Not completed — Death | 1
Period: At 3 Years Follow-up
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Started | 29
Completed | 28
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: At 4 Years Follow-up
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Started | 28
Completed | 23
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Death | 1
Period: At 5 Years Follow-up
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Started | 23
Completed | 15
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Withdrawal because of other reasons | 5
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 52
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Mitral Regurgitation Severity
Description: All patients were screened and determined eligible by Investigators who utilized transthoracic echocardiograms (TTE) to determine MR severity grades based on the American Society of Echocardiology recommendations for the determination of native valvular regurgitation. MR severity was assessed by an independent Echocardiography Core Laboratory (ECL).
Time Frame: At baseline
Population: Of total 55 patients,for 1 patient Echocardiogram was not evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 54
Percentage of participants
  0+:None | 0.0
  1+:Mild | 0.0
  2+:Moderate | 5.6
  3+:Moderate-to-Severe | 38.9
  4+:Severe | 55.6

2. Primary Outcome: Mitral Regurgitation Severity
Description: as for outcome 1
Time Frame: At discharge or within 30 days of the procedure
Population: Based on the number of patients who have not died or withdrawn, and have reached the scheduled visit window
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 48
Percentage of participants
  0+:None | 0.0
  1+:Mild | 62.5
  2+:Moderate | 20.8
  3+:Moderate-to-Severe | 14.6
  4+:Severe | 2.1

3. Primary Outcome: Mitral Regurgitation Severity
Description: as for outcome 1
Time Frame: At 12 months
Population: Of total 55 patients population 39 patients were analyzed, as for 1 patient Echocardiogram was not performed and 15 patients were withdrawn or lost to follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 39
Percentage of participants
  0+:None | 0.0
  1+:Mild | 35.9
  2+:Moderate | 35.9
  3+:Moderate-to-Severe | 17.9
  4+:Severe | 10.3

4. Primary Outcome: Mitral Regurgitation Severity
Description: as for outcome 1
Time Frame: At 24 months
Population: Of total 55 patients population 28 patients were analysed, as for 1 patient Echocardiogram was not performed and 15 patients were withdrawn or lost to follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 28
Percentage of participants
  0+:None | 0.0
  1+:Mild | 42.9
  2+:Moderate | 42.9
  3+:Moderate-to-Severe | 7.1
  4+:Severe | 7.1

5. Primary Outcome: Mitral Regurgitation Severity
Description: as for outcome 1
Time Frame: At 3 years
Population: Of total 55 patients population 23 patients were analysed, as for 5 patients Echocardiogram was not performed and 27 patients were withdrawn or lost to follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 23
Percentage of participants
  0+:None | 0.0
  1+:Mild | 39.1
  2+:Moderate | 39.1
  3+:Moderate-to-Severe | 13
  4+:Severe | 8.7

6. Primary Outcome: Mitral Regurgitation Severity
Description: as for outcome 1
Time Frame: At 4 years
Population: Of total 55 patients population 19 patients were analysed, as for 4 patients Echocardiogram was not performed and 32 patients were withdrawn or lost to follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 19
Percentage of participants
  0+:None | 0.0
  1+:Mild | 26.3
  2+:Moderate | 47.4
  3+:Moderate-to-Severe | 21.1
  4+:Severe | 5.3

7. Primary Outcome: Mitral Regurgitation Severity
Description: as for outcome 1
Time Frame: At 5 years
Population: Of total 55 patients population 15 patients were analysed, as 40 patients were withdrawn or lost to follow-up.
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 15
Percentage of participants
  0+:None | 0.0
  1+:Mild | 26.7
  2+:Moderate | 46.7
  3+:Moderate-to-Severe | 26.7
  4+:Severe | 0.0

8. Primary Outcome: Major Adverse Events (MAE)
Description: Defined in the Protocol as a combined clinical endpoint of death, myocardial infarction, cardiac tamponade, cardiac surgery for failed MitraClip device, single leaflet device attachment, stroke and septicemia.
Time Frame: Through 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants
  Death | 0
  Myocardial Infarction | 0
  Cardiac Tamponade | 1.8
  Cardiac Surgery for failed MitraClip Device | 1.8
  Single Leaflet Device Attachment (SLDA) | 7.2
  Stroke | 3.6
  Septicemia | 0

9. Primary Outcome: Major Adverse Events (MAE)
Description: as for outcome 8
Time Frame: Through 6 Months
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants
  Death | 1.8
  Myocardial Infarction | 1.8
  Cardiac Tamponade | 1.8
  Cardiac Surgery for failed MitraClip Device | 1.8
  Single Leaflet Device Attachment (SLDA) | 7.2
  Stroke | 3.6
  Septicemia | 1.8

10. Secondary Outcome: Procedure Time
Description: Procedure Time, defined as the time of start of the transseptal procedure to the time the Steerable Guide Catheter (SOC) is removed, averaged 255 minutes, or just over 4 hours.
  The reported Procedure Time includes the time required to collect Protocol required hemodynamic data pre- and post-implantation of the MitraClip device.
Time Frame: At day 0 (on the day of index procedure)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Minutes | 254.7 (105.1)

11. Secondary Outcome: Device Time
Description: Device Time, defined as the time of insertion of the Steerable Guide Catheter (SGC) to the time the MitraClip Delivery Catheter is retracted into the SGC.
Time Frame: At day 0 (on the day of index procedure)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Minutes | 198.5 (99.2)

12. Secondary Outcome: Contrast Volume
Description: Mean contrast volume utilized during the MitraClip procedure.
Time Frame: At day 0 (on the day of index procedure)
Population: Contrast volume was not recorded in one patient. Therefore, contrast volume data is available for 54 of the 55 patients.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 54
Milliliters | 112.0 (54.8)

13. Secondary Outcome: Fluoroscopy Duration
Description: Mean fluoroscopy duration during the MitraClip procedure.
Time Frame: At day 0 (on the day of index procedure)
Population: Mean fluoroscopy duration was not recorded in one patient. Therefore, mean fluoroscopy data is available for 54 of the 55 patients.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 54
Minutes | 59.8 (31.4)

14. Secondary Outcome: Number of Mitraclip Devices Implanted
Time Frame: At day 0 (on the day of index procedure)
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants
  0 | 10.9
  1 | 61.8
  2 | 27.3

15. Secondary Outcome: Intra-procedural Major Adverse Events
Description: Significant intra-procedural Major adverse events are defined as Major Adverse Events that occurred on the day of the procedure
Time Frame: At day 0 (on the day of index procedure)
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
percentage of participants
  Death | 0.0
  Myocardial Infarction | 0.0
  Cardiac Tamponade | 1.8
  Cardiac Surgery for failed MitraClip Device | 0.0
  Single Leaflet Device Attachment (SLDA) | 0.0
  Stroke | 1.8
  Septicemia | 0.0

16. Secondary Outcome: Post-procedure Intensive Care Unit (ICU)/Critical Care Unit (CCU)/Post-anesthesia Care Unit (PACU) Duration
Time Frame: Post index procedure within 30 days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Hours | 56.7 (80.2)

17. Secondary Outcome: Post-procedure Hospital Stay
Time Frame: Post-index procedure until hospital discharge (1 to 19 days)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Days | 2.9 (3.5)

18. Secondary Outcome: Second Intervention to Place a Second MitraClip Device
Time Frame: Post index procedure through 5 years
Measure: Number; unit: Participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Participants | 2

19. Secondary Outcome: MitraClip Device Embolizations and Single Leaflet Device Attachment
Description: MitraClip device embolizations means the detachment from both mitral leaflets. Single Leaflet Device Attachment (SLDA) is defined as the attachment of a single leaflet to the MitraClip device.
Time Frame: Post index procedure through 5 years
Population: Of the 55 patients enrolled in the EVEREST I study, 6 patients did not have a MitraClip device implanted.
Measure: Number; unit: Participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 49
Participants
  MitraClip device embolizations | 0
  Single Leaflet Device Attachment | 5

20. Secondary Outcome: Mitral Valve Surgery Post-MitraClip Device Implant Procedure (Kaplan-Meier Freedom From Mitral Valve Surgery)
Description: Freedom from mitral valve surgery required to treat mitral regurgitation and/or mitral stenosis and/or for Cardiac Surgery for Failed Clip following the MitraClip device procedure.
Time Frame: At baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 100

21. Secondary Outcome: Mitral Valve Surgery Post-MitraClip Device Implant Procedure (Kaplan-Meier Freedom From Mitral Valve Surgery)
Description: as for outcome 20
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 74.4 [60.28 to 84.11]

22. Secondary Outcome: Mitral Valve Surgery Post-MitraClip Device Implant Procedure (Kaplan-Meier Freedom From Mitral Valve Surgery)
Description: as for outcome 20
Time Frame: At 24 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 68.2 [52.25 to 79.75]

23. Secondary Outcome: Mitral Valve Surgery Post-MitraClip Device Implant Procedure (Kaplan-Meier Freedom From Mitral Valve Surgery)
Description: as for outcome 20
Time Frame: At 3 Years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 63.6 [47.65 to 75.88]

24. Secondary Outcome: Mitral Valve Surgery Post-MitraClip Device Implant Procedure (Kaplan-Meier Freedom From Mitral Valve Surgery)
Description: as for outcome 20
Time Frame: At 4 Years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 61.2 [44.58 to 74.16]

25. Secondary Outcome: Mitral Valve Surgery Post-MitraClip Device Implant Procedure (Kaplan-Meier Freedom From Mitral Valve Surgery)
Description: as for outcome 20
Time Frame: At 5 Years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 55.1 [34.86 to 71.32]

26. Secondary Outcome: Death (Kaplan-Meier Freedom From Death)
Time Frame: Within 30 days of the procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 100

27. Secondary Outcome: Death (Kaplan-Meier Freedom From Death)
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 97.7 [83.52 to 99.71]

28. Secondary Outcome: Death (Kaplan-Meier Freedom From Death)
Time Frame: At 24 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 95 [78.35 to 98.93]

29. Secondary Outcome: Death (Kaplan-Meier Freedom From Death)
Time Frame: At 3 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 95 [77.28 to 98.99]

30. Secondary Outcome: Death (Kaplan-Meier Freedom From Death)
Time Frame: At 4 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 91.5 [72.49 to 97.57]

31. Secondary Outcome: Death (Kaplan-Meier Freedom From Death)
Time Frame: At 5 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
Percentage of participants | 86.4 [59.22 to 96.01]

32. Secondary Outcome: Major Vascular and Bleeding Complications
Description: Major bleeding complications is defined as transfusion of >=2 units of blood due to bleeding related to the index procedure
Time Frame: Through 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
percentage of participants
  Major Vascular Complication | 5.5
  Major Bleeding Complication | 5.5
  Non-Cerebral Thromboembolism | 0.0

33. Secondary Outcome: Major Vascular and Bleeding Complications
Description: as for outcome 32
Time Frame: Through 6 Months
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
percentage of participants
  Major Vascular Complication | 7.3
  Major Bleeding Complication | 5.5
  Non-Cerebral Thromboembolism | 0.0

34. Secondary Outcome: Other Secondary Safety Events
Description: Other safety event includes Endocarditis, MitraClip DeviceThrombosis, Hemolysis, Mitral Valve Injury (major).
Time Frame: Through 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
percentage of participants
  Endocarditis | 0.0
  MitraClip Device Thrombosis | 0.0
  Hemolysis | 0.0
  Mitral Valve Injury (major) | 3.6

35. Secondary Outcome: Other Secondary Safety Events
Description: Other safety event includes Endocarditis, MitraClip DeviceThrombosis, Hemolysis, Mitral Valve Injury (major).
Time Frame: Through 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
percentage of participants
  Endocarditis | 1.8
  MitraClip Device Thrombosis | 0.0
  Hemolysis | 0.0
  Mitral Valve Injury (major) | 3.6

36. Secondary Outcome: Left Ventricular End Diastolic Volume
Description: Left Ventricular end-diastolic volume (LVEDV) as determined by the core echo laboratory. Left Ventricular end-diastolic volume (LVEDV) measured using 2-dimensional echocardiography. The endocardium is traced at end-diastole (frame before mitral valve closure or maximum cavity dimension) in the 2- and 4-chamber views to calculate volumes.
Time Frame: Baseline
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 51
Milliliter | 169.0 [157.3 to 180.7]

37. Secondary Outcome: Left Ventricular End Diastolic Volume
Description: as for outcome 36
Time Frame: During the hospital stay with a maximum of 3 days post index procedure (Discharge)
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 49
Milliliter | 154.8 [143.7 to 165.8]

38. Secondary Outcome: Left Ventricular End Diastolic Volume
Description: as for outcome 36
Time Frame: 12 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 39
Milliliter | 149.9 [137.8 to 161.9]

39. Secondary Outcome: Left Ventricular End Diastolic Volume
Description: as for outcome 36
Time Frame: 24 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 28
Milliliter | 131.4 [118.3 to 144.6]

40. Secondary Outcome: Left Ventricular End Diastolic Volume
Description: as for outcome 36
Time Frame: 60 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 9
Milliliter | 107.0 [82.2 to 131.8]

41. Secondary Outcome: Left Ventricular End Systolic Volume
Description: Left Ventricular end-systolic volume (LVESV) as determined by the core echo laboratory. Left Ventricular end-systolic volume (LVESV) measured using 2-dimensional echocardiography. The endocardium is traced at end-systole (frame prior to mitral valve opening or the minimum cavity area) in the 2- and 4-chamber views to calculate volumes.
Time Frame: Baseline
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 51
Milliliter | 67.0 [59.5 to 74.4]

42. Secondary Outcome: Left Ventricular End Systolic Volume
Description: as for outcome 41
Time Frame: During the hospital stay with a maximum of 3 days post index procedure (Discharge)
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 49
Milliliter | 67.4 [59.5 to 75.4]

43. Secondary Outcome: Left Ventricular End Systolic Volume
Description: Left Ventricular end-systolic volume (LVESV) as determined by the core echo laboratory. Left Ventricular end-systolic volume (LVESV) as determined by the core echo laboratory. Left Ventricular end-systolic volume (LVESV) measured using 2-dimensional echocardiography. The endocardium is traced at end-systole (frame prior to mitral valve opening or the minimum cavity area) in the 2- and 4-chamber views to calculate volumes.
Time Frame: 12 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 39
Milliliter | 62.8 [54.0 to 71.6]

44. Secondary Outcome: Left Ventricular End Systolic Volume
Description: as for outcome 43
Time Frame: 24 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 28
Milliliter | 55.8 [48.1 to 63.5]

45. Secondary Outcome: Left Ventricular End Systolic Volume
Description: as for outcome 43
Time Frame: 60 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 9
Milliliter | 40.4 [30.5 to 50.3]

46. Secondary Outcome: Mitral Valve Area - Single Orifice
Description: Mitral valve area measured by planimetry. Using a cineloop acquired at the mitral valve leaflet tips, the point in diastole corresponding to the maximal opening is identified. The area pre-device as well as post-device are planimetered. Post-device, the mitral valve orifice area is the sum of the area of each of the two orifices.
Time Frame: Baseline
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 47
cm^2 | 6.1 [5.7 to 6.6]

47. Secondary Outcome: Mitral Valve Area - Single Orifice
Description: as for outcome 46
Time Frame: During the hospital stay with a maximum of 3 days post index procedure (Discharge)
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 39
cm^2 | 3.7 [3.3 to 4.2]

48. Secondary Outcome: Mitral Valve Area - Single Orifice
Description: as for outcome 46
Time Frame: 12 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 32
cm^2 | 3.6 [3.1 to 4.0]

49. Secondary Outcome: Mitral Valve Area - Single Orifice
Description: as for outcome 46
Time Frame: 24 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 20
cm^2 | 3.4 [3.1 to 3.8]

50. Secondary Outcome: Mitral Valve Area - Single Orifice
Description: as for outcome 46
Time Frame: 60 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 5
cm^2 | 3.3 [2.3 to 4.3]

51. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-Time
Description: The pressure half time (PHT) measurement for assessing the severity of mitral stenosis is a widely accepted echocardiographic method.
  The decline of the velocity of diastolic transmitral blood flow is inversely proportional to mitral valve area (MVA), and MVA is derived using the empirical formula: MVA (cm^2) = 220/PHT PHT is calculated automatically by tracing the deceleration slope of the E-wave of transmitral flow, obtained with continuous wave Doppler echocardiography.
Time Frame: Baseline
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 43
cm^2 | 4.2 [3.9 to 4.5]

52. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-Time
Description: as for outcome 51
Time Frame: During the hospital stay with a maximum of 3 days post index procedure (Discharge)
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 40
cm^2 | 3.0 [2.6 to 3.3]

53. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-Time
Description: as for outcome 51
Time Frame: 12 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 39
cm^2 | 2.7 [2.5 to 3.0]

54. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-Time
Description: as for outcome 51
Time Frame: 24 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 28
cm^2 | 2.8 [2.5 to 3.2]

55. Secondary Outcome: Mitral Valve Area (MVA) by Pressure Half-Time
Description: as for outcome 51
Time Frame: 60 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 10
cm^2 | 2.8 [2.3 to 3.2]

56. Secondary Outcome: Mitral Valve Gradient
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: Baseline
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 47
mmHg | 1.7 [1.5 to 2.0]

57. Secondary Outcome: Mitral Valve Gradient
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: During the hospital stay with a maximum of 3 days post index procedure (Discharge)
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 47
mmHg | 3.9 [3.2 to 4.6]

58. Secondary Outcome: Mitral Valve Gradient
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 12 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 39
mmHg | 3.5 [3.0 to 4.0]

59. Secondary Outcome: Mitral Valve Gradient
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 24 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 28
mmHg | 3.7 [3.0 to 4.3]

60. Secondary Outcome: Mitral Valve Gradient
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by echocardiography.
Time Frame: 60 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 10
mmHg | 3.6 [2.8 to 4.3]

61. Secondary Outcome: Cardiac Output
Description: Cardiac output as measured by core lab echocardiography. Cardiac output is the product of forward stroke volume and heart rate.
Time Frame: Baseline
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 37
L/min | 3.7 [3.4 to 4.1]

62. Secondary Outcome: Cardiac Output
Description: as for outcome 61
Time Frame: During the hospital stay with a maximum of 3 days post index procedure (Discharge)
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 32
L/min | 4.7 [4.2 to 5.1]

63. Secondary Outcome: Cardiac Output
Description: as for outcome 61
Time Frame: 12 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 31
L/min | 4.2 [3.8 to 4.5]

64. Secondary Outcome: Cardiac Output
Description: as for outcome 61
Time Frame: 24 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 27
L/min | 4.2 [3.7 to 4.7]

65. Secondary Outcome: Cardiac Output
Description: as for outcome 61
Time Frame: 60 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 10
L/min | 3.7 [3.2 to 4.1]

66. Secondary Outcome: Cardiac Index
Description: Cardiac index is defined as cardiac output divided by body surface area. Cardiac Index is measured by core lab echocardiography.
Time Frame: Baseline
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min/m^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 34
L/min/m^2 | 2.0 [1.8 to 2.2]

67. Secondary Outcome: Cardiac Index
Description: as for outcome 66
Time Frame: During the hospital stay with a maximum of 3 days post index procedure (Discharge)
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min/m^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 29
L/min/m^2 | 2.5 [2.2 to 2.8]

68. Secondary Outcome: Cardiac Index
Description: as for outcome 66
Time Frame: 12 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min/m^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 27
L/min/m^2 | 2.2 [2.0 to 2.3]

69. Secondary Outcome: Cardiac Index
Description: as for outcome 66
Time Frame: 24 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min/m^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 23
L/min/m^2 | 2.3 [2.0 to 2.6]

70. Secondary Outcome: Cardiac Index
Description: as for outcome 66
Time Frame: 60 months
Population: Some patients are not analyzed due to non-evaluable echocardiograms or echocardiograms not done.
Measure: Mean (95% Confidence Interval); unit: L/min/m^2
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 10
L/min/m^2 | 2.1 [1.8 to 2.4]

71. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: Defined as assessment of NYHA functional class status at follow-up compared to baseline NYHA functional class status.
  Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 55
participants
  NYHA Functional Class I | 4
  NYHA Functional Class II | 24
  NYHA Functional Class III | 24
  NYHA Functional Class IV | 3

72. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 6 months
Population: NYHA functional class was evaluated in 41 patients at the 6-month follow-up visit. NYHA assessment is missing in 14 patients due to:
  * 7 withdrawals
  * 1 death
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 41
participants
  NYHA Functional Class I | 20
  NYHA Functional Class II | 17
  NYHA Functional Class III | 4
  NYHA Functional Class IV | 0

73. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 30 days
Population: NYHA functional class was evaluated in 47 patients at the 30-day follow-up visit. NYHA assessment is missing in 8 patients due to:
  * 2 withdrawals
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 47
participants
  NYHA Functional Class I | 27
  NYHA Functional Class II | 17
  NYHA Functional Class III | 3
  NYHA Functional Class IV | 0

74. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 12 months
Population: NYHA functional class was evaluated in 39 patients at the 12-month follow-up visit. NYHA assessment is missing in 16 patients due to:
  * 8 withdrawals
  * 1 death
  * NYHA assessment not done in 1 patient
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 39
participants
  NYHA Functional Class I | 19
  NYHA Functional Class II | 17
  NYHA Functional Class III | 3
  NYHA Functional Class IV | 0

75. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 18 months
Population: NYHA functional class was evaluated in 27 patients at the 18-month follow-up visit. NYHA assessment is missing in 28 patients due to:
  * 15 withdrawals
  * 2 deaths
  * 5 missed visits
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 27
participants
  NYHA Functional Class I | 15
  NYHA Functional Class II | 10
  NYHA Functional Class III | 1
  NYHA Functional Class IV | 1

76. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 24 months
Population: NYHA functional class was evaluated in 28 patients at the 24-month follow-up visit. NYHA assessment is missing in 27 patients due to:
  * 18 withdrawals
  * 2 deaths
  * 1 missed visit
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 28
participants
  NYHA Functional Class I | 15
  NYHA Functional Class II | 12
  NYHA Functional Class III | 1
  NYHA Functional Class IV | 0

77. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 36 months
Population: NYHA functional class was evaluated in 21 patients at the 36-month follow-up visit. NYHA assessment is missing in 34 patients due to:
  * 19 withdrawals
  * 2 deaths
  * 3 missed visits
  * 4 NYHA assessments not done
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 21
participants
  NYHA Functional Class I | 8
  NYHA Functional Class II | 10
  NYHA Functional Class III | 3
  NYHA Functional Class IV | 0

78. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 48 months
Population: NYHA functional class was evaluated in 19 patients at the 48-month follow-up visit. NYHA assessment is missing in 36 patients due to:
  * 23 withdrawals
  * 3 deaths
  * 1 missed visit
  * 3 NYHA assessments not done
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 19
participants
  NYHA Functional Class I | 6
  NYHA Functional Class II | 11
  NYHA Functional Class III | 2
  NYHA Functional Class IV | 0

79. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: as for outcome 71
Time Frame: 60 months
Population: NYHA functional class was evaluated in 15 patients at the 48-month follow-up visit. NYHA assessment is missing in 40 patients due to:
  * 30 withdrawals
  * 4 deaths
  * As per the protocol, the 6 patients not implanted with the MitraClip were not required to attend follow-up visits.
Measure: Number; unit: participants
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Number analyzed (Participants) | 15
participants
  NYHA Functional Class I | 5
  NYHA Functional Class II | 9
  NYHA Functional Class III | 1
  NYHA Functional Class IV | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Percutaneous Mitral Valve Repair (MitraClip Implant)
Serious Adverse Events (participants affected / at risk) | 36/55
Other Adverse Events (participants affected / at risk) | 43/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Percutaneous Mitral Valve Repair (MitraClip Implant) (N=55)
Anaemia (Blood and lymphatic system disorders) | 4
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 4
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 16
Myocardial infarction (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Death (General disorders) | 4
Mechanical complication of implant (General disorders) | 5
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Catheter sepsis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1
Device malfunction (Injury, poisoning and procedural complications) | 2
Bleeding time prolonged (Investigations) | 2
Haemoglobin decreased (Investigations) | 1
Urine output decreased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dementia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1
Blood product transfusion (Surgical and medical procedures) | 1
Cardiac operation (Surgical and medical procedures) | 1
Coronary revascularisation (Surgical and medical procedures) | 1
Hernia repair (Surgical and medical procedures) | 1
Hip surgery (Surgical and medical procedures) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Arteriovenous fistula (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Percutaneous Mitral Valve Repair (MitraClip Implant) (N=55)
Anaemia (Blood and lymphatic system disorders) | 5
Angina pectoris (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 8
Mitral valve incompetence (Cardiac disorders) | 8
Mitral valve stenosis (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 4
Chest pain (General disorders) | 5
Fatigue (General disorders) | 3
Injection site bruising (General disorders) | 3
Injection site haemorrhage (General disorders) | 22
Injection site pain (General disorders) | 8
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 5
Bleeding time prolonged (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 5
Orthostatic hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days